CLINICAL TRIAL: NCT00237081
Title: Maryland Genetics of Interstitial Cystitis (MaGIC)
Brief Title: Genetics of Interstitial Cystitis
Acronym: magic
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK66136-MaGIC (completed)
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2010-03

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: Interstitial Cystitis; Painful Bladder Syndrome; Genetics; Risk factors; Family history
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The cause of interstitial cystitis is unknown. However, it tends to run in some families suggesting that there may be a genetic susceptibility to the disease. For instance, the disease is found 17 times more commonly in first-degree relatives (parent, sibling, or child) of patients with interstitial cystitis than in the general population. Furthermore, if one twin has interstitial cystitis, the disease is much more common in identical co-twins than fraternal co-twins. This evidence suggests that, in some families, genes that make a person susceptible to interstitial cystitis are being passed from one generation to the next.

The University of Maryland School of Medicine and the National Institutes of Health are performing a study to identify these genes for susceptibility for interstitial cystitis. This study is entitled the Maryland Genetics of Interstitial Cystitis (MaGIC) study. The MaGIC study will investigate several hundred families with two or more blood relatives with interstitial cystitis. The study will seek to find changes in genes that are found far more commonly in family members who have interstitial cystitis than in those who do not have the disease.Identifying these genes should lead to a better understanding of the cause of interstitial cystitis. Finding the cause is the first step to finding the cure.

This is a national study which is conducted by telephone and mail, and in which you can participate entirely from your home.

ELIGIBILITY:
Inclusion Criteria:

* Have interstitial cystitis, or painful bladder syndrome.
* Have at least one blood relative with interstitial cystitis, painful bladder syndrome, or urinary symptoms similar to yours.
* Are 13 years of age or older.
* Are available for a telephone, mail, or website interview.
* Live in the USA or Canada.

Exclusion Criteria:

* Are less than 13 years of age.
* Have Parkinson's disease, Multiple Sclerosis, Spina bifida, or another neurologic disease that preceeded your interstitial cystitis symptoms

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-06; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Warren, M.D., Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Interstitial Cystitis Center, Baltimore, Maryland, United States

REFERENCES:
- See also: Interstitial Cystitis Association — http://www.ichelp.org
- See also: Interstitial Cystitis Network — http://www.ic-network.com